CLINICAL TRIAL: NCT04125576
Title: Comparison of Pain-Related Changes in Cerebral Blood Volume in Burn Patients With Neuropathic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: HangangSHH-5
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Neuropathic Pain
Keywords: burn; neuropathic pain; cerebral blood volume
MeSH Terms: conditions — Neuralgia; Burns | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Burn patients: The subjects complaine of severe neuropathic pain that is rated at least 5 on the visual analogue scale (VAS), despite treatments with gabapentin medication and other physical modalities.
  Interventions: Diagnostic Test: magnetic resonance imaging(MRI)
- Healthy controls: age and sex matched healthy controls
  Interventions: Diagnostic Test: magnetic resonance imaging(MRI)

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging(MRI) — magnetic resonance imaging(MRI) will be used to evaluate cerebral blood volume(CBV) of pain network

SUMMARY:
The investigators will observe increased or decreased CBV in patients with thermal injury compared with the CBV in healthy controls.

DETAILED DESCRIPTION:
Prevalence of chronic pain has been shown to be high after thermal injury. Post-burn neuropathic pain causes chronic disabilities that is often difficult to treat effectively.

To study changes in the pain network associated with neuropathic pain, magnetic resonance imaging(MRI) will be used to evaluate cerebral blood volume(CBV) in patients who was injuried by burn. Over the fifty participants will be recruited. The participants will be comprised 30 subjects with neuropathic pain caused by thermal injury and 20 healthy contols. The 30 patients with neuropathic pain will be comprised divided into 15 electrical injury group and 15 non-electrical burn injury group. The patients are included the patients with severe neuropathic pain that is rated at least 5 on the visual analogue scale (VAS), despite treatments with gabapentin medication and other physical modalities. The intensity of neuropathic pain will be measured using the visual analogue scale(VAS). Depressive mood will be assessed using the Beck Depression Scale. CBV maps will be compared between burn patients and controls. And the relationship between individual participant CBV(measured in voxels), BDS and VAS score will be also examined.

ELIGIBILITY:
Inclusion Criteria:

* Burn patients
* severe neuropatic pain rated at least 5 on the 10-point numerical rating scale (NRS).

Exclusion Criteria:

* cardiac arrest history
* history of neurologic disease or brain surgery
* unstable heart disease or presence of a cardiac pacemaker
* psychiatric disorder
* diabetes mellitus
* abnormal renal function
* contraindication for MRI
* pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patients complained of severe neuropatic pain rated at least 5 on the 10-point numerical rating scale (NRS), despite being treated with drugs and physical therapy for more than 1 week after being admitted to the Department of Rehabilitation Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
cerebral blood volume | 1 week
  magnetic resonance imaging(MRI) was used to evaluate cerebral blood volume(CBV) of pain network

SECONDARY OUTCOMES:
visual analogue scale | 1 week
  The intensity of neuropathic pain was measured using the visual analogue scale, Zero ("0") represented no pain and 10 represented unbearable symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park CH, Seo CH, Jung MH, Joo SY, Jang S, Lee HY, Ohn SH. Investigation of cognitive circuits using steady-state cerebral blood volume and diffusion tensor imaging in patients with mild cognitive impairment following electrical injury. Neuroradiology. 2017 Sep;59(9):915-921. doi: 10.1007/s00234-017-1876-1. Epub 2017 Jul 8. PMID 28689261
- [Background] Seo CH, Park CH, Jung MH, Jang S, Joo SY, Kang Y, Ohn SH. Preliminary Investigation of Pain-Related Changes in Cerebral Blood Volume in Patients With Phantom Limb Pain. Arch Phys Med Rehabil. 2017 Nov;98(11):2206-2212. doi: 10.1016/j.apmr.2017.03.010. Epub 2017 Apr 6. PMID 28392326